CLINICAL TRIAL: NCT01429025
Title: A Pilot/Feasibility Phase I Study of Bendamustine, Rituximab and Lenalidomide in Patients With Refractory/Relapsed Indolent NHL
Brief Title: Rituximab, Bendamustine Hydrochloride, and Lenalidomide in Treating Patients With Refractory or Relapsed Indolent Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N1088; NCCTG-N1088; CDR0000710726 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-03535 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Refractory/Relapsed Indolent Non-Hodgkin Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; Waldenström macroglobulinemia; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; Bendamustine Hydrochloride; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab, bendamustine and lenalidomide (Experimental): Patients receive rituximab IV on day 1, bendamustine IV on days 1-2, and lenalidomide PO on days 1-10. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: bendamustine; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — IV
Drug: bendamustine — IV
Drug: lenalidomide — PO

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as bendamustine hydrochloride, also work in different ways to kill cancer cells or stop them from dividing. Lenalidomide may stop the growth of non-Hodgkin lymphoma by blocking blood flow to the cancer. Giving lenalidomide together with rituximab and bendamustine hydrochloride may kill more cancer cells.

PURPOSE: This phase I trial studies the side effects and the best dose of giving lenalidomide together with rituximab and bendamustine hydrochloride in treating patients with refractory or relapsed indolent non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a pilot/feasibility study of bendamustine, rituximab, and lenalidomide combination with a goal of assessing maximum tolerated dose, safety and feasibility of this combination. Patients receive rituximab IV over 5-8 hours on day 1, bendamustine hydrochloride IV over 30-60 minutes on days 1-2, and lenalidomide orally (PO) on days 1-10. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Ancillary treatment is available per the protocol (eg, supportive care for rituximab infusions).

OBJECTIVES:

Primary

* To establish the maximum-tolerated dose of lenalidomide in combination with bendamustine and rituximab chemotherapy

Secondary

* To evaluate the toxicity profile of lenalidomide in combination with bendamustine and rituximab chemotherapy
* To assess progression-free survival
* To assess the overall and complete response rates of lenalidomide in combination with bendamustine and rituximab in patients with relapsed/refractory indolent non-Hodgkin lymphoma (NHL)

Patients may undergo blood sample collection at baseline and periodically during treatment for correlative studies. Tumor tissue samples may also be collected.Patients are followed up for up to 5 years post-registration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically confirmed relapsed (recurrent after previous therapy (-ies)) or refractory (no response to previous therapy (-ies)), CD20 + indolent/low-grade B-cell non-Hodgkin lymphoma (NHL) expressing CD20 antigen. Criteria for diagnosis can be found in reference J Clin Oncol 17(4): 1244-53, 1999. The biopsy confirming relapse can be up to 12 weeks prior to registration as long as there is no intervening therapy. If patients have been on active treatment within the the last 12 weeks, the tumor biopsy must be repeated before study enrollment to evaluate for transformation.

   * Small lymphocytic lymphoma (SLL) excluding chronic lymphocytic leukemia (CLL) (patients with peripheral blood lymphocyte count > 5,000)
   * Follicular lymphoma, grades 1, 2 (grade 3 excluded)
   * Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphatic tissue (MALT) type
   * Lymphoplasmacytic lymphoma including Waldenstrom macroglobulinemia
3. Measurable disease (at least 1 lesion of ≥ 1.5 cm in diameter) as detected by computed tomography (CT) or the CT images of the positron emission tomography (PET)/CT. Patients with Waldenstrom macroglobulinemia are not required to have measurable disease by CT or PET/CT if monoclonal protein is detectable by serum protein electrophoresis and/or IgM level is at least 2 times upper limit of normal
4. ECOG Performance Status (PS) 0, 1 or 2
5. Required laboratory values obtained ≤ 21 days prior to registration:

   * ANC ≥ 1,500/mL
   * Platelet count ≥ 100,000/mL
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) OR, if total bilirubin is > 1.5 x ULN, the direct bilirubin must be normal
   * SGOT (AST) ≤ 5 x ULN
   * Creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula as outlined in the protocol
6. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®. The Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods are provided in the protocol for more information.

   * Females of childbearing potential (FCBP) as defined per the protocol must have:

     1. A negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL ≤10 - 14 days prior to registration and again ≤ 24 hours prior to starting cycle 1 of lenalidomide
     2. ≥28 days prior to registration, throughout the duration of the study, and for up to 28 days from the last dose of lenalidomide, FCBP must agree to either continued abstinence from heterosexual intercourse or must begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME
     3. Must agree to ongoing pregnancy testing throughout the duration of the study and for up to 28 days from the last dose of lenalidomide.
   * Men must agree to abstinence or to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
7. Willing to provide informed written consent.
8. Willing to return to enrolling institution for follow-up.
9. If currently not on anticoagulation medication, willing and able to take low-dose aspirin (81 mg) daily. NOTE: The dose of aspirin should be a minimum of 81 mg and can be higher if the patient is on the agent for other reasons. If aspirin is contraindicated, the patient may be considered for the study after consultation with the study chair regarding other alternatives including the possible use of warfarin or low molecular weight heparin. Patients unable to take any prophylaxis are not eligible.
10. Life expectancy ≥6 months
11. Ability to swallow oral medications

Exclusion Criteria:

1. This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant women
   * Nursing women (lactating females are eligible provided that they agree not to breast feed while taking lenalidomide)
   * Men or women of childbearing potential who are unwilling to employ adequate contraception
2. Active CNS lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells that requires therapy
3. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
4. Prior AIDS-defining conditions. Note: HIV positive patients without history of AIDS- defining conditions are eligible

   * If HIV positive, CD4 cells < 400/mm^3
   * Current treatment with zidovudine (AZT) (which may cause overlapping adverse events, primarily myelosuppression). Patients receiving anti-retroviral therapy other than AZT are eligible
5. Uncontrolled intercurrent illness including, but not limited to:

   * Ongoing or active infection
   * Symptomatic congestive heart failure
   * Unstable angina pectoris
   * Cardiac arrhythmia
   * Psychiatric illness/social situations that would limit compliance with study requirements
6. Receiving any other agent which would be considered as a treatment for the lymphoma.

   Note: Prior use of rituximab is allowed.
7. Another active malignancy requiring concomitant active therapy such as radiation, chemotherapy, or immunotherapy. Exceptions to this are as follows:

   * Localized non-melanotic skin cancer
   * Cancers that are inactive that are being treated with hormonal therapy
   * Any cancer that in the judgment of the investigator will not interfere with the study treatment plan and response assessment and require concomitant anticancer therapy for the duration of this study

   Contact the study chair regarding any questions related to eligibility of patients with concomitant active malignancy
8. History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
9. History of life threatening (i.e. pulmonary embolism), DVT or recurrent thrombosis/embolism and are not on or unwilling to receive anticoagulation

   * Patients with history of DVT or life threatening or recurrent thrombosis/embolism (PE) may enter the study but must receive anticoagulation with low molecular weight (LMW) heparin or therapeutic warfarin during the protocol treatment and for ≥6 months afterwards. Patients with strong family history of thrombosis should be considered for thrombophilia work up and/or anticoagulated at the discretion of treating MD.
   * Patients with a prior history (>6 months prior to study entry) of a non-life threatening, provoked thrombosis (e.g. history of catheter related thrombus or similar) and without known thrombophilia can participate in the study and receive standard prophylaxis with ASA (aspirin) or LMW heparin/warfarin at the discretion of treating MD. Active smokers should be advised on thrombosis risk and smoking cessation and may participate in the study if prophylaxis with ASA (aspirin) or LMW heparin/warfarin (at the discretion of treating MD) is given. Patients on estrogen birth control pills should be advised of the risks.
10. Known myelodysplastic syndrome
11. Receiving erythroid stimulating agents (EPO: Procrit, Aranesp). Note: Use of erythroid stimulating agents is not allowed during the study treatment.
12. Prior treatment with bendamustine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of lenalidomide in combination with bendamustine hydrochloride and rituximab | Up to 28 days

SECONDARY OUTCOMES:
Toxicity profile | Up to 5 years
Progression-free survival | Time from registration to the earliest date of documented disease progression or death due to any cause, assessed up to 5 years
Overall response rate | Up to 5 years
Complete response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz S. Nowakowski, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (17):
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota